CLINICAL TRIAL: NCT03048240
Title: A Pilot Study of the Feasibility of Intraoperative Photodynamic Therapy of Glioblastoma.
Brief Title: INtraoperative photoDYnamic Therapy of GliOblastoma
Acronym: INDYGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016_06; 2016-002706-39 (EudraCT Number)
Record Dates: First submitted 2017-01-24; First posted 2017-02-09 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2020-11

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "perPDT" (Experimental): Single arm : per-operative PhotoDynamic Therapy (perPDT) during the surgery of Glioblastoma excision.
  Interventions: Device: "perPDT"; Drug: GLIOLAN

INTERVENTIONS:
Device: "perPDT" — The protocol requires the realization of specific procedures in addition to the usual care.
  The per-operative photodynamic therapy ("perPDT") added to surgery for glioblastoma excision. The patient will receive 5-ALA (5- alanine ,GLIOLAN drinkable) 4h before surgery + lighting of the tumor bed by a light source (laser) at the end of resection (Prolonged surgery of 45 minutes).
Drug: GLIOLAN — patient will receive 5-ALA (5- alanine ,GLIOLAN drinkable) 4h before surgery

SUMMARY:
The study pilot evaluate the feasibility of a "5-ALA- PpIX (protoporhyrin IX) mediated per-PDT protocol" in patients with glioblastoma accessible for complete surgical removal of contrast. This treatment will be carried out in addition to the current reference treatment of glioblastoma: maximum resection surgery followed by radiochemotherapy according to the protocol Stupp

ELIGIBILITY:
Inclusion Criteria:

1. Patient male or female ≥18 years
2. General status (WHO) of Performance status 0, 1 or 2
3. Probable glioblastoma according to clinical and radiological criteria,
4. whose surgical indication was given in Multidisciplinary consultation meeting (RCP) of neurooncology,
5. Decision to treat the patient as part of the Clinical trial also taken in neuro-oncology RCP ("Multidisciplinary consultation meeting")
6. Patient operable on the basis of absence of cardiopulmonary disease history; a complete medical check-up sufficient to insure a post-operative state with normal daily life
7. Clinical neuro-oncological monitoring and long-term MRI scheduled at the hospital CHRU of Lille, center of reference of the region
8. Patient able to understand and sign voluntarily Informed consent
9. Patient able to adhere to the visit's calendar of the study and other imperatives of the protocol
10. Women of child-bearing potential should benefit of an effective contraception
11. For patients receiving hepatotoxic therapy in the long term, this treatment must be suspended during the 24h after taking 5-ALA
12. Patient assigned to an heath insurance

Exclusion Criteria:

1. Contraindications to 5-ALA (Gliolan®) and to per-operative PhotoDynamic Therapy "perPDT":
2. Contraindications to 5-ALA

   * Porphyria
   * Taking photosensitizer treatment
   * Severe renal or hepatic impairment
   * Bilirubin> 1.5 x maximum level, Alkaline Phosphatases and transaminases (ASAT)> 2.5 x Maximum. rates
   * Creatinine clearance <30 mL / min;
   * Non-compliance with the rules of prevention of the transient risk of cutaneous photosensitization
3. Contraindications to surgery
4. Contraindications to magnetic resonance imaging (MRI)
5. Treatment with an experimental drug within 30 Days prior to the start of the study
6. Clinical follow-up impossible to perform for psychological, familial, social or geographical reasons,
7. Legal incapacity (persons deprived of their liberty or Guardianship or guardianship),
8. Pregnant or nursing women
9. Refusal to participate or sign the consent of the study
10. Soy allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Number of Patients having the full "PerPDT" treatment with unacceptable and unexpected toxicities (grade ≥ 3) graded According to NCI CTC Version 4.0 | From the intake of Gliolan (5-Ala) until 1 month post "perPDT"
  In particular, the following complications will be investigated: severe infection, new neurological deficit responsible for severe disability, status epilepticus, deaths during the postoperative period.
  Target: At least 6/10 patients who benefited of complete "PerPDT" and without unacceptable and unexpected toxicities

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From the Date of diagnosis of glioblastoma until the date of Relapse defined, assessed up to 24 months
  Determined according to international RANO criteria
Overall Survival (OS) | From the date of Diagnosis of glioblastoma until the date of death, assessed up to 24 months
  Determined according to international RANO criteria
Response to treatment | From the date of perPDT until relapse/death, assessed up to 24 months
  Evaluated by MRI every 3 months
Incidence of "per PDT" treatment-emergent Adverse Events | From the beginning of treatment with perPDT up to relapsing/death, assessed up to 24 months
  Collection of all Adverse events (AEs and SAEs) (according to NCI-CTC V4.0) and reviewing by an Independent Safety Monitoring Board.
Quality of Life Questionnaire -C30 ( QLQ-C30) | Every 3 months from the signature of Consent form until relapse/death, assessed up to 24 months
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
Quality of Life Questionnaire - Brain Cancer Module (QLQ-BN20) | Every 3 months from the signature of Consent form until relapse/death, assessed up to 24 months
  Measuring the health-related quality of life in patients with brain cancer

OTHER OUTCOMES:
Analyze of Peripheral Blood Mononuclear Cells | Every 3 months from the signature of Consent form until relapse/death, assessed up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Reyns, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vermandel M, Dupont C, Lecomte F, Leroy HA, Tuleasca C, Mordon S, Hadjipanayis CG, Reyns N. Standardized intraoperative 5-ALA photodynamic therapy for newly diagnosed glioblastoma patients: a preliminary analysis of the INDYGO clinical trial. J Neurooncol. 2021 May;152(3):501-514. doi: 10.1007/s11060-021-03718-6. Epub 2021 Mar 20. PMID 33743128
- [Derived] Peciu-Florianu I, Vannod-Michel Q, Vauleon E, Bonneterre ME, Reyns N. Long term follow-up of patients with newly diagnosed glioblastoma treated by intraoperative photodynamic therapy: an update from the INDYGO trial (NCT03048240). J Neurooncol. 2024 Jul;168(3):495-505. doi: 10.1007/s11060-024-04693-4. Epub 2024 May 16. PMID 38753093